CLINICAL TRIAL: NCT04956068
Title: Pressurized Intra-Peritoneal Aerosol Chemotherapy (PIPAC) for Peritoneal Metastases
Brief Title: PIPAC for Peritoneal Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC
Record Dates: First submitted 2021-05-24; First posted 2021-07-09 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Peritoneal Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unresectable PM group (Experimental): Patients who have progressed on conventional systemic therapy and PIPAC is used as a palliative strategy.
  Interventions: Combination Product: PIPAC
- Extensive PM group (Experimental): Patients who have significant volume of peritoneal disease are treated with the intent for potential conversion to curative surgery. Role of PIPAC is as an adjunct to systemic chemotherapy to downstage peritoneal metastases.
  Interventions: Combination Product: PIPAC

INTERVENTIONS:
Combination Product: PIPAC — A novel drug delivery system using the CapnoPen device which allows the aerolisation of chemotherapeutic agents within the peritoneal cavity. PIPAC procedure will be carried out with either oxaliplatin or doxorubicin/ cisplatin.

SUMMARY:
Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a novel drug delivery system that allows the direct application of chemotherapeutic agents into the peritoneal cavity. It boosts improved distribution, enhanced tissue uptake and repeatability using minimally invasive access. It was devised to palliate the local symptoms of extensive peritoneal metastases (PM) in patients who are not amenable to curative surgery. This study is to determine safety and feasibility of PIPAC in patients with PM from Gastrointestinal (GI) cancer, Hepato-Pancreato-Biliary (HPB) cancer, and other rare malignancies.

ELIGIBILITY:
Inclusion Criteria:

For Unesectable PM Group:

* Age ≥ 21 years old
* ECOG < 3
* Fit for systemic chemotherapy treatment
* Adequate bone marrow function (haemoglobin ≥ 8.0 mmol/L, neutrophils ≥ 1.5X109/L, platelets ≥ 100X109/L
* Adequate renal function (e-GFR > 30mls/min for patients undergoing PIPAC with oxaliplatin; e-GFR > 60mls/min for patients undergoing PIPAC with Doxorubicine/Cisplatin)
* Adequate liver function (Total bilirubin < 1.5 upper limit of normal; ALT and AST< 3 upper limit of normal)
* No contraindications to chemotherapy agents oxaliplatin, doxorubicin/ cisplatin
* No contraindications to general anaesthesia and diagnostic laproscopy procedure
* Normal left ventricular ejection fraction (for patients undergoing PIPAC with doxorubicin/ cisplatin)
* Histological/ cytological proof of PM from GI, HPB, Gynaecology, Breast, Sarcoma primaries
* Peritoneal-dominant metastatic disease

For the Extensive PM Group:

All the above mentioned criteria as for the unresectable group, with the addition of the following:

* Not suitable for curative cytoreductive surgery (CRS) & hyperthermic intraperitoneal chemotherapy (HIPEC) surgery after diagnostic laproscopy - PCI > 18 in LGI, PCI > 6 in UGI ECOG < 3
* In UGI PM patients, progression while on bidirectional chemotherapy

Exclusion Criteria:

* Patient is medically unfit for surgery due to concurrent medical comorbidities, including but not limited to intestinal obstruction, multiple sites of metastases
* Any medical or psychiatric condition(s) which would preclude informed consent
* Patient is pregnant or nursing
* GI PM patients with PCI >6 but are treatment naive (these patients should undergo standard treatment - bidirectional intravenous and intraperitoneal chemotherapy)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with major toxicities of at least CTCAE Grade 3 and above | Up to 4 weeks after each PIPAC procedure
  To determine and safety and feasibility of PIPAC in patients with PM. Common Terminology Criteria for Adverse Events (CTCAE) measures Grade 1 to 5, with higher grade indicating greater severity.
Number of patients with minor toxicities of CTCAE Grade 1 and 2 | Up to 4 weeks after each PIPAC procedure
  Common Terminology Criteria for Adverse Events (CTCAE) measures Grade 1 to 5, with higher grade indicating greater severity.
Length of hospitalisation stay for each PIPAC procedure | Through study completion, an average of half a year

SECONDARY OUTCOMES:
Intra-operative Peritoneal Carcinomatosis Index (PCI) score | During each PIPAC procedure
  To examine the clinical response of PM after PIPAC. PCI score from 0 to 39 with a higher number representing a greater amount of disease present in the peritoneum.
Ascites volume | During each PIPAC procedure
  To examine the clinical response of PM after PIPAC
Peritoneal Regression Grading Score (PRGS) from PM biopsy | At each PIPAC procedure
  To examine the clinical response of PM after PIPAC
Quality of Life Assessment using Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire | At 4 time points - Baseline (before any PIPAC procedure), pre-2nd PIPAC (Before 2nd PIPAC procedure), pre-3rd PIPAC (before 3rd PIPAC procedure) and 4 weeks post-3rd PIPAC (4 weeks after 3rd PIPAC procedure)
  Range: 0-108. A high score represents a better health state
Quality of Life Assessment using European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Quality of life questionnaire | At 4 time points - Baseline (before any PIPAC procedure), pre-2nd PIPAC (Before 2nd PIPAC procedure), pre-3rd PIPAC (before 3rd PIPAC procedure) and 4 weeks post-3rd PIPAC (4 weeks after 3rd PIPAC procedure)
  Range: 0-100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Progression free survival | From the start of the first PIPAC procedure, up to 5 years
Overall survival | From the start of the first PIPAC procedure, up to 5 years
Percentage of patients that convert to curative surgery | From the start of the first PIPAC procedure, up to 24 weeks ± 4 weeks
  (Only applicable for Extensive PM group)

CONTACTS AND LOCATIONS:
Overall Officials: Claramae Chia, MBBS, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No